CLINICAL TRIAL: NCT02336906
Title: A Controlled Randomized, Physician Blinded Study to Assess Isolated Uro-therapy vs. Urotherapy With Constipation Treatment for Patients With Lower Urinary Tract Dysfunction (LUTD) Not Meeting ROME-III Constipation Criteria
Brief Title: Urotherapy vs. Urotherapy With Constipation Treatment for Children With Lower Urinary Tract Dysfunction
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Changes in departmental staff have led to a cut in research alotments.
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Noam Zevit, Pediatric Gastroenterologist, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rmc130348ctil
Record Dates: First submitted 2015-01-01; First posted 2015-01-13 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Diurnal Enuresis
Keywords: Lower urinary tract dysfunction; constipation
MeSH Terms: conditions — Diurnal Enuresis; Constipation | interventions — polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urotherapy + Constipation Treatment (Active Comparator): This group will be treated with standard behavioral urotherapy in addition to receiving active stool softening with PEG3350 and standard constipation instruction.
  Interventions: Drug: polyethylene glycol 3350; Behavioral: Constipation behavioral therapy; Behavioral: Urotherapy
- Urotherapy alone (Other): This group will receive standard behavioral urotherapy alone.
  Interventions: Behavioral: Urotherapy

INTERVENTIONS:
Drug: polyethylene glycol 3350 — Patients will initially receive three days of high dose PEG3350 treatment (1.5gr/kg up to 100gr maximum) and the stepped down to 0.8gr/kg subsequently tapered according to stool consistency and frequency.
  Other Names: PEG3350; Normalax
  Arms: Urotherapy + Constipation Treatment
Behavioral: Constipation behavioral therapy — Patients in the active group will receive dietary instruction as to fiber content, as well as behavior therapy including active sitting on the toilet to attempt defacation following meals.
  Arms: Urotherapy + Constipation Treatment
Behavioral: Urotherapy — The children will be guided for appropriate drinking and toilet habits, and will start with timed voiding.

SUMMARY:
Constipation treatment has been found to ameliorate symptoms in some patients with lower urinary tract dysfunction (including day time or combined day time/night time urinary incontinence). This study aims to explore if treatment of patients without overt constipation (As defined by the ROME III criteria) will also respond to anti-constipation treatment with reduction of their urinary tract symptoms. Assessment of severity and response of lower urinary tract dysfunction will be based on the Vancouver NULTD/DES questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 5-17 years at time of signing of informed consent.
2. Lower urinary tract dysfunction (LUTD)-daytime/daytime and nighttime urinary incontinence as defined by a score of >11 on the Vancouver Questionnaire .
3. Do not meet Rome III criteria for functional constipation.

Exclusion Criteria:

1. Inability to provide signed informed consent.
2. Inability to comply with the study protocol.
3. Neurogenic bladder
4. Attention Deficit Disorder (ADD or ADHD) on medical treatment.
5. Known significant sacral, perineal, or other congenital or surgical defect.
6. Known orthopedic/neurological disease which may affect urinary continence, cause constipation, or affect reading of abdominal x-rays. (e.g. spastic cerebral palsy, severe scoliosis)
7. Patient taking medicinal drugs which can cause urinary incontinence or constipation.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Complete (Vancouver score - ≤90% of screening value) or Partial (Vancouver score ≤ 50% screening value) response at the end of intervention. | 14 weeks

SECONDARY OUTCOMES:
Number of participants with complete (Vancouver score - ≤90% of screening value) or Partial (Vancouver score ≤ 50% screening value) response in patient subgroups with fecal loading compared to those without fecal loading. | 14 weeks
  Number of participants with complete (Vancouver score - ≤90% of screening value) or Partial (Vancouver score ≤ 50% screening value) response to therapy in those with radiological evidence of fecal loading on enrollment abdominal x-ray (as defined by rectal/pelvic outlet ratio, Leech score, and Barr score) compared to those who did not in the intervention group and the urotherapy group
Sustained Response - Number of participants with complete (Vancouver score - ≤90% of screening value) or Partial (Vancouver score ≤ 50% screening value) response 12 weeks after intervention has ended. | 26 weeks
Number of participants with adverse effects | 14 weeks
  Adverse effects of interventions as reported by patients/care givers during visits

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Gastroenterology, Nutrition, and Liver Diseases; Schneider Children's Medical Center of Israel, Petah Tikva, Israel

REFERENCES:
- [Background] Afshar K, Mirbagheri A, Scott H, MacNeily AE. Development of a symptom score for dysfunctional elimination syndrome. J Urol. 2009 Oct;182(4 Suppl):1939-43. doi: 10.1016/j.juro.2009.03.009. Epub 2009 Aug 20. PMID 19695637
- [Background] Hodges SJ, Anthony EY. Occult megarectum--a commonly unrecognized cause of enuresis. Urology. 2012 Feb;79(2):421-4. doi: 10.1016/j.urology.2011.10.015. Epub 2011 Dec 14. PMID 22173180